CLINICAL TRIAL: NCT07210996
Title: A Single-center, Open-label, Randomized, Single Dose, Two-way Crossover Design to Evaluate the Relative Bioavailability of Pimicotinib Capsules Containing Free Base in Different Proportions Under Fasting Conditions in Healthy Participants
Brief Title: A Study to Evaluate the Relative Bioavailability of Pimicotinib Capsules Containing Free Base in Different Proportions in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ABSK021-113
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pharmacokinetics in Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pimicotinib (test capsule-reference capsule) (Other): subjects in sequence A will receive a single oral dose of 50 mg test capsule administered as 2 x 25 mg (free base content at certain level) in period 1 day 1 and receive a single oral dose of 50 mg reference capsule administered as 2 x 25 mg (free base content below detection limit) in period 2 day 1.
  Interventions: Drug: pimicotinib capsules
- pimicotinib (reference capsule-test capsule) (Other): subjects in sequence B will receive a single oral dose of 50 mg reference capsule administered as 2 x 25 mg ((free base content below detection limit) in period 1 day 1 and receive a single oral dose of 50 mg test capsule administered as 2 x 25 mg (free base content at certain level) in period 2 day 1 .
  Interventions: Drug: pimicotinib capsules

INTERVENTIONS:
Drug: pimicotinib capsules — pimicotinib capsules

SUMMARY:
This is an open-label, randomized, two-treatment, single-dose, two-way crossover study to evaluate the relative bioavailability and tolerability of Pimicotinib capsules containing free base in different proportions in healthy participants. 20 healthy participants are planned to be enrolled and will be evenly randomized to either Study Sequence A or Study Sequence B.Subjects in Sequence A/Sequence B will receive a single 50 mg oral dose of test/reference pimicotinib in period 1 and cross over in period 2. Blood samples will be collected for PK analysis in totally 32 time-points.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants aged 18 to 50 years (inclusive) at screening and at least 25% of each sex should be included.
2. Weight ≥ 50.0 kg (male) or ≥ 45.0 kg (female), with a body mass index (BMI) between 18 and 28 (inclusive), BMI = weight (kg)/height (m)2;
3. Normal or abnormal but not clinically significant results in medical history, physical examination, clinical laboratory tests and other relevant examinations as assessed by the investigator at Screening;
4. Male or female participants of childbearing potential must agree to use effective methods of contraception during the study and within 6 months after the last dose of investigational product , and male participants should not donate sperm during such period; female participants should not donate ovum during such period and should not be pregnant or lactating. Pregnancy period is defined as the period from the date of conception until termination of pregnancy, and will be determined by laboratory test of human chorionic gonadotropin (hCG) within 7 days prior to initiation of the study;
5. Willing to participate in this study, understand the study procedures and sign the informed consent form prior to screening; willing to comply with the study procedures.

   -

Exclusion Criteria:

1. Past or current medical history of chronic or severe conditions in cardiovascular, respiratory, blood, liver, kidney, gastrointestinal, endocrine or nervous systems;
2. Known or persistent mental disorders that may preclude the subject from participation in the study, as determined by the investigator;
3. Past history of gastric or intestinal surgery, or other operations (except for appendectomy) affecting the drug absorption;
4. Dysphagia and inability to take the investigational product orally;
5. Intolerant to venipuncture, difficult to collect blood samples, and fear of needle sickness and blood;
6. Known allergy to two or more kinds of foods and drugs; or allergic to pimicotinib or its excipients (lactose monohydrate, microcrystalline cellulose, colloidal silicon dioxide, croscarmellose sodium, magnesium stearate, gelatin); and prone to allergic reactions such as rash and urticaria;
7. History of bacterial, fungal, parasitic, viral (excluding nasopharyngitis), mycobacterial infection, and COVID-19 infection within 30 days prior to screening; or abnormal chest X-ray (posteroanterior view) finding, assessed as clinically significant (by the investigator);
8. Symptoms of fatigue and pyrexia within 2 weeks prior to screening;
9. Abnormal laboratory tests: Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) > 1.2 × Upper Limit of Normal (ULN); Creatinine > 1.2 × ULN; Total Bilirubin (TBIL) > 1.5 × ULN; Creatine Kinase (CK) > 1.5 × ULN and amylase > 1.2 × ULN; hemoglobin <115g/L for Male or < 105g/L for Female;
10. Positive result for either of the following tests: serum Hepatitis B Surface Antigen (HBsAg), Hepatitis C Virus (HCV) antibody, Human Immunodeficiency Virus (HIV) antibody, and treponema pallidum antibody;
11. Participated in any clinical studies of drugs as a study subject and received the study drug within 3 months prior to screening;
12. Previously participated in any other study related to pimicotinib and received pimicotinib;
13. Used strong inhibitors or inducers of CYP3A4 within 14 days prior to screening and at Screening or intending to use during the study;
14. Have special diet requirements and cannot accept to take a unified dietary; specific dietary requirements the participants can only eat the food provided by the study site during hospitalization;
15. Consumption of more than 14 units of alcohol per week within 3 months prior to signing the informed consent form, or a positive result for alcohol breath test on the day pre-dose, or unable to abstain from alcohol during the study;
16. Consumption of more than 5 cigarettes per day within 3 months prior to signing the informed consent form, or unable to abstain from tobacco products during the study;
17. Previous chronic consumption of excessive amount of tea, coffee, or caffeinated beverages or unable to abstain from caffeinated beverages during the study;
18. Known history of drug abuse or positive for drug abuse screening test ;
19. Used over the counter or prescription drugs, including herbal medicine, health products, vitamins, and dietary supplements, within 14 days prior to screening, or plan to use such drugs during the study;
20. Donated or lost > 400 mL of blood within 3 months prior to screening; received blood transfusions or used blood products within 2 months prior to screening;
21. Received vaccine (including COVID-19 vaccine) within 2 months prior to screening, or plan to get vaccinated during the study;
22. Significant abnormalities and judged by the investigator as clinical significance in vital signs, including: forehead temperature > 37.6 °C; pulse rate > 100 beats/min or < 50 beats/min; systolic blood pressure ≥ 140 mmHg, diastolic blood pressure ≥ 90 mmHg;
23. Heart rate-corrected QT interval prolongation, QTcF > 470 ms (> 480 ms for females) (Note: QTc interval corrected using the Fridericia formula), or family history of long QT syndrome, or other clinically significant ECG abnormalities at Screening;
24. Participants involved in the design or conduct of this study and their immediate family members;
25. Participants who, in the opinion of the investigator, are not suitable for enrollment or may not be able to complete the study for other reasons.

    -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-09-12 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Cmax | Period 1& Period 2: pre-dose, postdose 15 minutes, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 24 hours, 48 hours, 96 hours, 120 hours, 144 hours, 192 hours and 240 hours.
  Peak concentration, the maximum observed plasma concentration of pimicotinib
AUC0-∞ | Period 1& Period 2: pre-dose, postdose 15 minutes, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 24 hours, 48 hours, 96 hours, 120 hours, 144 hours, 192 hours and 240 hours.
  Area under the plasma concentration-time curve of pimicotinib from time 0 to infinity, calculated as: AUC0-∞=AUClast +Clast/λz; Clast refers to the last measurable (non-BQL) plasma concentration of pimicotinib
AUClast | Period 1& Period 2: pre-dose, postdose 15 minutes, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 24 hours, 48 hours, 96 hours, 120 hours, 144 hours, 192 hours and 240 hours.
  Area under the plasma concentration-time curve of pimicotinib from time 0 to the time of last measurable (non-BQL) concentration (calculated using the Linear Up Log Down trapezoidal method)

SECONDARY OUTCOMES:
AE | through study completion, an average of 26 days
  To evaluate the safety following a single oral dose of the two different pimicotinib capsules under fasting conditions in healthy subjects,The relationship of each adverse event to the investigational product will be assessed by CTCAE v5.0.
t1/2 | Period 1& Period 2: pre-dose, postdose 15 minutes, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 24 hours, 48 hours, 96 hours, 120 hours, 144 hours, 192 hours and 240 hours.
  Elimination half-life
CL/F | Period 1& Period 2: pre-dose, postdose 15 minutes, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 24 hours, 48 hours, 96 hours, 120 hours, 144 hours, 192 hours and 240 hours
  Total apparent clearance after a single oral dose
Vz/F | Period 1& Period 2: pre-dose, postdose 15 minutes, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 24 hours, 48 hours, 96 hours, 120 hours, 144 hours, 192 hours and 240 hours
  Apparent volume of distribution after a single oral dose

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojiao Li, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No